CLINICAL TRIAL: NCT03951857
Title: Biphasic and Combined Effect of Aging & Obesity With Development of Effective Exercise Intervention Protocol
Brief Title: Effect of Aging & Obesity With Exercise Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Jae-Young Lim, Professor, Department of Rehabilitation Medicine, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B-1610-365-001
Record Dates: First submitted 2019-05-10; First posted 2019-05-15 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Obesity
Keywords: Aging; Obesity; Single muscle fiber contractile properties; Intramyocellular lipids; Resistance exercise
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Young men (No Intervention): Range of age is 20-35 years, young men (BMI 19-23 Kg/m2) They did not suffer from musculoskeletal or metabolic diseases, and had not performed regular exercise within the previous 3 months.
- Young women (No Intervention): Range of age is 20-35 years, young women (BMI 19-23 Kg/m2) They did not suffer from musculoskeletal or metabolic diseases, and had not performed regular exercise within the previous 3 months.
- Elderly women (control) (Experimental): Range of age is 65-80 years, Elderly women (BMI 19-23 Kg/m2) They did not suffer from musculoskeletal or metabolic diseases, and had not performed regular exercise within the previous 3 months.
  Interventions: Other: Resistance exercise with a gym stick
- Elderly obese women (Experimental): Range of age is 65-80 years,Elderly obese women (BMI ≥25 Kg/m2) They did not suffer from musculoskeletal or metabolic diseases, and had not performed regular exercise within the previous 3 months.
  Interventions: Other: Resistance exercise with a gym stick

INTERVENTIONS:
Other: Resistance exercise with a gym stick — Exercise intervention: The resistance exercise intervention is performed with a gym stick for 3 times a week for 12 weeks. Exercise load is gradually increased by the number of times the band is wound and the speed of motion by dividing into three stages in 1-4 weeks (1st stage), 5-8 weeks (2nd stage) and 9-12 weeks (3rd stage).
  Other Names: Exercise training
  Arms: Elderly obese women; Elderly women (control)

SUMMARY:
Obesity leads to a vicious circle that increases intramuscular fat, insulin resistance, promotes muscular dysfunction resulting in increased muscle fat accumulation. The study of muscle function and intramyocellular lipids is insufficient for obesity. Particularly, the study of mechanisms in muscle function and intramyocellular lipids is few nationally and internationally.

DETAILED DESCRIPTION:
This study is prospective study. The goal of this study is

1. To examine the distribution and contractile properties (cross-sectional area, maximal force, specific force, maximal shortening velocity) of single muscle fiber sex/Myosin heavy chain (MHC) type-related differences, by extracting a single muscle fiber from the vastus lateralis in young men and women.
2. To examine the effects of intramyocellular lipids on physical activity ability, muscle dysfunction, and metabolic disorders in relation to aging and obesity.
3. To examine the effects of intramyocellular lipids on physical activity ability, muscular dysfunction, and metabolic disorders after 12 weeks resistance exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Young men: Age (20-35 yrs), BMI (19-23 Kg/m2)
* Young women: Age (20-35 yrs), BMI (19-23 Kg/m2)
* Elderly women: Age (65-80 yrs), BMI (19-23 Kg/m2)
* Elderly obese women: Age (65-80 yrs), BMI ( >25 Kg/m2)
* Subjects who can agree voluntarily.

Exclusion Criteria:

* Acute coronary syndrome.
* Uncontrolled hypertension.
* Subjects who took drugs which can affects neuromuscular system.
* Severely impaired cognition
* Subjects who cannot agree voluntarily

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is divided into two purposes.
  1. To examine the distribution and contractile properties (CSA, Po, SF, Vo) of single muscle fiber sex/MHC type-related differences in youn men and women.
  2. To examine effects of 12-week resistance exercise on single muscle fiber funtion and intramyocellular lipids in aging and obese elderly women.
  For the purposes of the first study, young men and women (age 20-35 yrs) should be participated in this study.
  aimed to examine the distribution and contractile properties (CSA, Po, SF, Vo) of single muscle fiber sex/MHC type-related differences, by extracting a single muscle fiber from the vastus lateralis in young men and women
Enrollment: 28 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Total droplet area | Before intervention / after 12weeks intervention
  Change from baseline total droplet area to 12 weeks after initial assessment. Total droplet area is determined by Oil-red-O staining. After staining, the total area (µm2) is analyzed to compare the change after intervention from baseline.
Number of lipid droplets | Before intervention / after 12weeks intervention
  Change from baseline number of lipid droplets to 12 weeks after initial assessment.
  Number of lipid droplets determined by Oil-red-O staining. After staining, number of lipid droplets is analyzed to compare the change after intervention from baseline.
Single muscle fiber cross-sectional area (CSA) | Before intervention / after 12weeks intervention
  Change from baseline CSA to 12 weeks after initial assessment. Chemically skinned vastus lateralis muscle fiber CSA (µm2) is measured by 3 dimensional microscopy. after analysis, CSA is compared the change after intervention from baseline.
Single muscle fiber maximal force (Po) | Before intervention / after 12weeks intervention
  Change from baseline Po to 12 weeks after initial assessment. Chemically skinned vastus lateralis muscle fiber Po (mN) is measured by slack test procedure. after measurement, Po is analyzed to compare the change after intervention from baseline.
Single muscle fiber specific force (SF) | Before intervention / after 12weeks intervention
  Change from baseline SF to 12 weeks after initial assessment. Chemically skinned vastus lateralis muscle fiber SF (kN/m2) is Po (kN) normalized by cross-sectional area (m2). SF is analyzed to compare the change after intervention from baseline.
Single muscle fiber maximal shortening velocity (Vo) | Before intervention / after 12weeks intervention
  Change from baseline Vo to 12 weeks after initial assessment. Chemically skinned vastus lateralis muscle fiber Vo (FL/s) is measured by slack test procedure. The time required to take up the imposed slack was measured from the onset of the length step to the beginning of the tension redevelopment . For each amplitude of length, the ﬁber was reextended while relaxed to minimize nonuniformity of sarcomere length. A straight line was presented to a plot of length vs. time, using least-squares regression, and the slope of the line divided by the segment length was recorded as Vo for that ﬁber.
  Vo is analyzed to compare the change after intervention from baseline.
Single muscle fiber MHC type distribution | Before intervention / after 12weeks intervention
  Change from baseline fiber type distribution to 12 weeks after initial assessment.
  The MHC composition of single fibers was determined by sodium dodecyl sulfate-polyacrylamide gel electrophoresis (SDS-PAGE).
  MHC type distribution is analyzed to compare the change after intervention from baseline.

SECONDARY OUTCOMES:
Hand grip strength | Before intervention / after 12weeks intervention
  Change from baseline hand grip strength to 12 weeks after initial assessment. Participants are tested while they were seated, their arms are against their sides, their elbows are flexed 90 degrees. Hand grip Strength is measured in kilograms (kg) using a hand-grip dynamometer. The maximum value from either hand is used for analysis.
Isokinetic knee extension strength | Before intervention / after 12weeks intervention
  Change from baseline Knee extension strength to 12 weeks after initial assessment.
  Isokinetic knee extension strength is measured in as peak torque achieved on an isokinetic dynamometer (BTE Primus, BTE tech, MD, USA) at 60° per second.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Youn Lim, Ph.D., Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lexell J, Taylor CC, Sjostrom M. What is the cause of the ageing atrophy? Total number, size and proportion of different fiber types studied in whole vastus lateralis muscle from 15- to 83-year-old men. J Neurol Sci. 1988 Apr;84(2-3):275-94. doi: 10.1016/0022-510x(88)90132-3. PMID 3379447
- [Background] Doherty TJ, Vandervoort AA, Brown WF. Effects of ageing on the motor unit: a brief review. Can J Appl Physiol. 1993 Dec;18(4):331-58. doi: 10.1139/h93-029. PMID 8275048
- [Background] Goodpaster BH, Park SW, Harris TB, Kritchevsky SB, Nevitt M, Schwartz AV, Simonsick EM, Tylavsky FA, Visser M, Newman AB. The loss of skeletal muscle strength, mass, and quality in older adults: the health, aging and body composition study. J Gerontol A Biol Sci Med Sci. 2006 Oct;61(10):1059-64. doi: 10.1093/gerona/61.10.1059. PMID 17077199
- [Background] Hughes VA, Frontera WR, Wood M, Evans WJ, Dallal GE, Roubenoff R, Fiatarone Singh MA. Longitudinal muscle strength changes in older adults: influence of muscle mass, physical activity, and health. J Gerontol A Biol Sci Med Sci. 2001 May;56(5):B209-17. doi: 10.1093/gerona/56.5.b209. PMID 11320101
- [Background] Goodpaster BH, Krishnaswami S, Resnick H, Kelley DE, Haggerty C, Harris TB, Schwartz AV, Kritchevsky S, Newman AB. Association between regional adipose tissue distribution and both type 2 diabetes and impaired glucose tolerance in elderly men and women. Diabetes Care. 2003 Feb;26(2):372-9. doi: 10.2337/diacare.26.2.372. PMID 12547865
- [Background] Tuttle LJ, Sinacore DR, Mueller MJ. Intermuscular adipose tissue is muscle specific and associated with poor functional performance. J Aging Res. 2012;2012:172957. doi: 10.1155/2012/172957. Epub 2012 May 14. PMID 22666591
- [Background] Yim JE, Heshka S, Albu J, Heymsfield S, Kuznia P, Harris T, Gallagher D. Intermuscular adipose tissue rivals visceral adipose tissue in independent associations with cardiovascular risk. Int J Obes (Lond). 2007 Sep;31(9):1400-5. doi: 10.1038/sj.ijo.0803621. Epub 2007 Apr 24. PMID 17452994
- [Background] Visser M, Kritchevsky SB, Goodpaster BH, Newman AB, Nevitt M, Stamm E, Harris TB. Leg muscle mass and composition in relation to lower extremity performance in men and women aged 70 to 79: the health, aging and body composition study. J Am Geriatr Soc. 2002 May;50(5):897-904. doi: 10.1046/j.1532-5415.2002.50217.x. PMID 12028178
- [Background] Koster A, Ding J, Stenholm S, Caserotti P, Houston DK, Nicklas BJ, You T, Lee JS, Visser M, Newman AB, Schwartz AV, Cauley JA, Tylavsky FA, Goodpaster BH, Kritchevsky SB, Harris TB; Health ABC study. Does the amount of fat mass predict age-related loss of lean mass, muscle strength, and muscle quality in older adults? J Gerontol A Biol Sci Med Sci. 2011 Aug;66(8):888-95. doi: 10.1093/gerona/glr070. Epub 2011 May 13. PMID 21572082
- [Background] Addison O, Marcus RL, Lastayo PC, Ryan AS. Intermuscular fat: a review of the consequences and causes. Int J Endocrinol. 2014;2014:309570. doi: 10.1155/2014/309570. Epub 2014 Jan 8. PMID 24527032
- [Background] Goodpaster BH, Carlson CL, Visser M, Kelley DE, Scherzinger A, Harris TB, Stamm E, Newman AB. Attenuation of skeletal muscle and strength in the elderly: The Health ABC Study. J Appl Physiol (1985). 2001 Jun;90(6):2157-65. doi: 10.1152/jappl.2001.90.6.2157. PMID 11356778
- [Background] Yoshida Y, Marcus RL, Lastayo PC. Intramuscular adipose tissue and central activation in older adults. Muscle Nerve. 2012 Nov;46(5):813-6. doi: 10.1002/mus.23506. PMID 23055318
- [Background] Visser M, Goodpaster BH, Kritchevsky SB, Newman AB, Nevitt M, Rubin SM, Simonsick EM, Harris TB. Muscle mass, muscle strength, and muscle fat infiltration as predictors of incident mobility limitations in well-functioning older persons. J Gerontol A Biol Sci Med Sci. 2005 Mar;60(3):324-33. doi: 10.1093/gerona/60.3.324. PMID 15860469
- [Background] Ryan AS, Ortmeyer HK, Sorkin JD. Exercise with calorie restriction improves insulin sensitivity and glycogen synthase activity in obese postmenopausal women with impaired glucose tolerance. Am J Physiol Endocrinol Metab. 2012 Jan 1;302(1):E145-52. doi: 10.1152/ajpendo.00618.2010. Epub 2011 Oct 18. PMID 22008454
- [Background] Santanasto AJ, Glynn NW, Newman MA, Taylor CA, Brooks MM, Goodpaster BH, Newman AB. Impact of weight loss on physical function with changes in strength, muscle mass, and muscle fat infiltration in overweight to moderately obese older adults: a randomized clinical trial. J Obes. 2011;2011:516576. doi: 10.1155/2011/516576. Epub 2010 Oct 10. PMID 20953373
- [Background] Gorgey AS, Mather KJ, Cupp HR, Gater DR. Effects of resistance training on adiposity and metabolism after spinal cord injury. Med Sci Sports Exerc. 2012 Jan;44(1):165-74. doi: 10.1249/MSS.0b013e31822672aa. PMID 21659900
- [Background] Menshikova EV, Ritov VB, Fairfull L, Ferrell RE, Kelley DE, Goodpaster BH. Effects of exercise on mitochondrial content and function in aging human skeletal muscle. J Gerontol A Biol Sci Med Sci. 2006 Jun;61(6):534-40. doi: 10.1093/gerona/61.6.534. PMID 16799133
- [Background] Choi SJ, Files DC, Zhang T, Wang ZM, Messi ML, Gregory H, Stone J, Lyles MF, Dhar S, Marsh AP, Nicklas BJ, Delbono O. Intramyocellular Lipid and Impaired Myofiber Contraction in Normal Weight and Obese Older Adults. J Gerontol A Biol Sci Med Sci. 2016 Apr;71(4):557-64. doi: 10.1093/gerona/glv169. Epub 2015 Sep 23. PMID 26405061